CLINICAL TRIAL: NCT05393557
Title: Upfront Premedication For Reduction of Microvascular Obstruction and No-reflow in Treating ST-segment Elevation Myocardial Infarction
Acronym: UPFRONT-STEMI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Aswan Heart Centre (Other)
Responsible Party: Principal Investigator, Ahmad Samir, MD, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20220204MYFAHC
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: STEMI; Large Thrombus Burden; No-Reflow Phenomenon
Keywords: No reflow; STEMI; Glycoprotein inhibitor; repeated intermittent balloon inflation; reperfusion injury
MeSH Terms: conditions — ST Elevation Myocardial Infarction; No-Reflow Phenomenon; Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Upfront (Active Comparator): Immediately after restoration of distal flow, they will receive:
  i. Small dose Tirofiban (intra-coronary bolus of 25µg/Kg),[22] ii. Nitroglycerin 100-200 µg,[12] iii. Verapamil 100-200 µg (excluding patients with 2nd or 3rd degree AV block, bradycardia HR < 60, or systolic BP <100 mmHg)[5] iv. Two cycles of balloon up-balloon down (15 seconds occlusion, 15 seconds open artery; repeated two times).
  v. The rest of the procedure will be completed as standard practice.
  Interventions: Other: Upfront preparation of microcirculation to minimize risks of no-reflow and reperfusion injury
- Control (No Intervention): pPCI procedure will be performed as per standard practice.[2] Bail-out use of any pharmaceutical products will be allowed as per guidelines recommendations (such as: GPi in case of no-reflow or thrombotic complications).

INTERVENTIONS:
Other: Upfront preparation of microcirculation to minimize risks of no-reflow and reperfusion injury — Tirofiban (intra-coronary bolus of 25µg/Kg) + Nitroglycerin (intracoronary 100-200 µg) + Verapamil (intracoronary 100-200 µg, yet excluding patients with 2nd or 3rd degree AV block, HR < 60, or SBP <100 mmHg) + 2 cycles of intermittent balloon inflation
  Arms: Upfront

SUMMARY:
Angiographic no-reflow during primary PCI procedures occurs at relatively high rate (25%) and is associated with worsening of long term morbidity and mortality. The exact mechanism of no-reflow is not fully understood, yet it is believed to be multifactorial including microvascular plugging with activated platelets and thrombotic debris in addition to the microvascular dysfunction from the ischaemia-reperfusion injury.

Despite a theoretical advantage of glycoprotein IIb/IIIa inhibitors (GPi) (like; Tirofiban) to suppress the intense platelets' activation/reaction; their use did not lead to a significant net benefit, because it was opposed by increased risk of bleeding.

However, the bleeding that plagued GPi use was predominantly related to vascular access in the era femoral approach was the default. Moreover, there are some recent data suggesting that small intracoronary bolus of GPi was non-inferior to intravenous bolus-infusion dose with less bleeding events.

This study plans to assess upfront premedication with small doses of GPi + Nitroglycerin ± Verapamil, with staged restoration of flow (repeated balloon inflation) to reduce angiographic no-reflow and CMR assessed microvascular occlusion (MVO).

DETAILED DESCRIPTION:
A. Study Design This study will be a randomized single blinded prospective study including acute STEMI patients presenting to Aswan heart centre catheterization-lab for pPCI. All patients will undergo pPCI according to the current practice guidelines[1,2] and the local hospital policy in managing STEMI patients.

B. Study Population Acute STEMI patients presenting for pPCI reperfusion (or recuse PCI), identified upon initial wiring of the IRA to have large thrombus burden (TIMI thrombus grade 4-5).

C. Study Site This study with all planned diagnostic and therapeutic protocol will be performed in Aswan Heart Centre, Magdi Yacoub Foundation.

D. Study Protocol

1. Patients identified to have large thrombus burden (TIMI-thrombus grade 4 and 5), will be assigned into one of two groups according to a closed envelope randomization system.
2. Group A (active arm);

Immediately after restoration of distal flow, they will receive:

i. Small dose Tirofiban (intra-coronary bolus of 25µg/Kg),[22] ii. Nitroglycerin 100-200 µg,[12] iii. Verapamil 100-200 µg (excluding patients with 2nd or 3rd degree AV block, bradycardia HR < 60, or systolic BP <100 mmHg)[5] iv. Two cycles of balloon up-balloon down (15 seconds occlusion, 15 seconds open artery; repeated two times).

v. The rest of the procedure will be completed as standard practice. c. Group B (control arm); pPCI procedure will be performed as per standard practice.[2] Bail-out use of any pharmaceutical products will be allowed as per guidelines recommendations (such as: GPi in case of no-reflow or thrombotic complications).

d. Patients' baseline data will be collected on site using a standardized case report form directly into a web-based research data collection tool (REDCAP). Baseline characteristics, medical history, biochemical and electrocardiographic findings, prior chronic therapies and treatments administered during hospitalization will be comprehensively tabulated. On admission, blood samples will be collected from all patients to perform routine labs (CBC, INR, renal function test and serum electrolytes), hs-troponin-I, BNP and hs-CRP, according to institutional practice. An initial bed-side echo targeting assessment of LV dimensions and systolic function, significant valvular dysfunction, and exclusion mechanical complications will be performed without delay of revascularization.

e. After procedure completion, the following parameters will be collected: i. Occurrence of slow flow/no reflow after stent deployment or stent optimization (TIMI flow < 3) ii. Final TIMI flow iii. Final corrected TIMI flow count iv. Final TIMI myocardial blush grade v. Final TIMI myocardial perfusion grade vi. ST segment resolution assessed immediately (within 30 minutes). ST segment resolution will be quantified both in the index lead and as sum of the affected leads.

vii. Peak cardiac troponin within 24 hours of presentation. viii. Hemoglobin drop (baseline - lowest hemoglobin value during the hospital stay), overt bleeding, need for blood products transfusion will be collected. Bleeding events will be classified according to BARC categories as follows: Type 1: is bleeding that "is not actionable" and does not cause the patient to seek medical attention. Type 2: includes any clinically overt sign of hemorrhage that "is actionable" and requires diagnostic studies, hospitalization, or treatment by a healthcare professional. Type 3 has 3 subdivisions. Type 3a bleeding includes any transfusion with overt bleeding and overt bleeding plus a hemoglobin drop of ≥3 to <5 g/dL (provided the hemoglobin drop is related to bleeding). Type 3b bleeding includes overt bleeding plus a hemoglobin drop of ≥5 g/dL (provided the hemoglobin drop is related to bleeding), cardiac tamponade, bleeding requiring surgical intervention for control (excluding dental/nasal/skin/hemorrhoid), and bleeding requiring intravenous vasoactive drugs. Type 3c bleeding includes intracranial hemorrhage and intraocular bleeding compromising vision. Type 4 bleeding is coronary artery bypass grafting (CABG)-related (within 48 hours), and type 5 bleeding is fatal which should be categorized as intracranial, gastrointestinal, retroperitoneal, pulmonary, pericardial, or genitourinary.

ix. All patients will receive guidelines directed medical therapy as appropriate [2], and will receive similar advice for the required secondary preventive life-style changes.

x. A comprehensive echocardiographic and CMR examination will be performed predischarge (within 48 hours from presentation) to serve as baseline assessment.

xi. At 90-days post procedure, patients will have a mandatory clinical visit for clinical, echocardiographic and CMR follow-up assessment.

E. Potential Risks:

Primary PCI is considered the gold-standard therapy and is highly recommended to be timely performed in all patients presenting by acute STEMI. Potential risks for pPCI procedures include coronary dissection, perforation, procedural failure, significant bleeding complications or procedural related mortality, however, these complications are very rare (<1%) and substantially counterbalanced by the procedural benefits on short- and long terms. Active group receiving small doses of (GPi) are theoretically at increased risk for bleeding, which is mitigated by giving small dose. Also, committing the study eligibility to radial access only will further reduce the bleeding risk substantially, because radial access in pPCI was reported to reduce the bleeding risk to the half, compared to femoral access.[2]

F. Confidentiality of data:

Clinical data will be tabulated by number codes that will be anonymized. Only treating physicians will have access to participants identities, while the anonymized tabulated data will be available for the steering committee and the statisticians.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients with time from symptom onset of < 24 hours duration.
* Large thrombus burden confirmed after initial wiring.
* Radial vascular access.

Exclusion Criteria:

* STEMI patients receiving successful fibrinolytic therapy.
* TIMI flow ≥ 1 or TIMI thrombus grade ≤ 3 at initial wiring.
* Refusal to participate int the study, or unable to be consented (unconscious or comatose patients).
* Femoral access.
* Previous infarction in the same territory.
* Patients receiving PTCA only for acute reperfusion and planned for CABG.
* Patients with known intolerance or contraindications for CMR, such as claustrophobic or those with mechanical heart valve prothesis, or implantable non-conditional heart rhythm devices.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint: Reducing rates of suboptimal PCI results | One day (assessed by the end of the procedure)
  Sub-optimal PCI results defined as any of:
  1. Final TIMI flow < 3, TIMI myocardial blush grade < 3, corrected TIMI flow count (cTFC) < 20,
  2. Occurrence of TIMI flow < 3 during stenting/post dilation, (no reflow)
  3. ST elevation resolution < 50% in the index lead assessed within 30m from the procedural end.
Safety endpoint: Occurrence of intrahospital BARC types 3 or 5 bleedings | 30 days
  Occurrence of intrahospital BARC types 3 or 5 bleedings

SECONDARY OUTCOMES:
Occurrence of slow flow/no reflow after stent deployment or stent optimization (TIMI flow < 3) | one day (assessed by the end of the procedure)
  occurrence of TIMI flow < 3 after stent deployment or post stent optimization
Final TIMI flow | one day (assessed by the end of the procedure)
  TIMI flow at the end of the procedure
Final TIMI myocardial blush grade | One day (assessed by the end of the procedure)
  TIMI myocardial blush grade at the end of the procedure
NT-BNP at 90 days | 90 days
  N-terminal pro brain natriuretic peptide
LVEF at 90 days | 90 days
  Left ventricular ejection fraction
MVO at 90 days assessed by CMR | 90 days
  Microvascular obstruction assessed by cardiac magnetic resonance assessed by 90 days
Myocardial salvage assessed by CMR | 90 days
  Comparing infarction size at 90 days to area at risk (AAR) in baseline CMR study
Adverse remodeling of the LV | 90 days
  Increase of LVEDV and LVESV by ≥ 12% in the 90-days CMR from baseline .

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Samir, Principal Investigator — Aswan Heart Centre